CLINICAL TRIAL: NCT04202497
Title: A Phase 1, Open-label, Positron Emission Tomography Study With [18F]MNI-1054 to Determine Lysine-Specific Demethylase 1A Brain Enzyme Occupancy of TAK-418 After Single-Dose Oral Administration in Healthy Subjects
Brief Title: A Study With [18F]MNI-1054 to Determine Lysine -Specific Demethylase 1A (LSD1) Brain Enzyme Occupancy of TAK-418 After Single-Dose Oral Administration in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was prematurely terminated because of administrative reasons.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-418-0004; U1111-1242-8485 (Registry Identifier: WHO)
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — TAK-418

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-418 1.5 mg (Experimental): TAK-418 1.5 milligram (mg), orally, once on Day 1. Participants will also receive 10 millicurie (mCi) of [18F]MNI-1054 injection intravenously, prior to each PET scans on Day -1, Day 1, and either on Day 2 or 3. Dose levels for subsequent participants may vary based on available review of imaging and pharmacokinetics (PK) data.
  Interventions: Drug: TAK-418; Drug: [18F]MNI-1054 (radiotracer)

INTERVENTIONS:
Drug: TAK-418 — TAK-418 orally.
Drug: [18F]MNI-1054 (radiotracer) — [18F]MNI-1054 injection.

SUMMARY:
The purpose of this study is to determine brain LSD1 enzyme occupancy and the relationship of occupancy to TAK-418 dose and plasma exposure after single oral dosing of TAK-418 in healthy participants using [18F]MNI-1054 positron emission tomography (PET) imaging.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-418. TAK-418 is being tested to determine the relationship between brain LSD1 enzyme occupancy and TAK-418 plasma concentration. This study will utilize the PET radiotracer [18F]MNI-1054 to evaluate the brain LSD1 enzyme occupancy of TAK-418 after single dose oral administration in healthy adult participants.

The study will enroll approximately 16 participants. The TAK-418 starting dose is 1.5 mg, given on Day 1. Each participant will receive one dose of TAK-418 and up to 3 dynamic [18F]MNI-1054 PET scans to assess enzyme occupancy on baseline, Day 1 and Day 2 or 3 post-TAK-418 dosing.

This single center trial will be conducted in the United States. The overall time to participate in this study is 62 days. Participants will be followed up on Day 14 for follow-up safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must have a body mass index (BMI) greater than or equal to (>=) 18.5 and less than or equal to (<=) 30.0 kilogram per square meter (kg/m^2) at the screening visit.
2. The participant must be a current nonsmoker at screening as demonstrated by negative cotinine test.
3. The participant has adequate circulation to both hands for safe placement of arterial lines (as determined by Allen's test).

Exclusion Criteria:

1. Has a known hypersensitivity to any component of the formulation of TAK-418 or related compounds, including [18F]MNI-1054.
2. The participant has a positive alcohol or drug screen.
3. The participant has a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to the following: beer [354 milliliter (mL)/12 ounce (oz)], wine [118 mL/4 oz], or distilled spirits [29.5 mL/1 oz] per day).
4. The participant consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
5. The participant has a substance abuse disorder.
6. The participant cannot tolerate venipuncture or has poor venous access that would cause difficulty in collecting blood samples.
7. The participant has contraindications to undergoing magnetic resonance imaging (MRI) examination including but not limited to implants, such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, central nervous system aneurysm clips, and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.
8. The participant has clinically significant abnormal findings on brain MRI scan that in the opinion of the investigator may interfere with the interpretation of the PET imaging.
9. The participant has experienced an acute illness within 10 days before the screening visit.
10. The participant has a risk of suicide according to the investigator's clinical judgement per the Columbia-Suicide Severity Rating Scale at screening or has made a suicide attempt in the 12 months before screening.
11. The participant has luteinizing hormone, follicle stimulating hormone (FSH), or estradiol levels that are clinically abnormal.
12. The participant has existing skin rashes that can be diagnosed as dermatitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Invicro, A Konica Minolta Company, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 18 December 2019 to 19 March 2020.
Pre-assignment Details: Healthy participants were enrolled in this study to receive up to 10 millicurie [mCi]) of [18F]MNI-1054 for 1 positron emission tomography (PET) Scan on Day -1 (Baseline Scan), and then eligible participants entered into 1 of 3 treatment groups in the Treatment Period to receive 10 mCi of [18F]MNI-1054 for 2 PET scans after single dose of TAK-418 1.5 milligram (mg), 10 mg, or 30 mg on Day 1 and either Day 2 or 3. Study was prematurely terminated because of administrative reasons.
Groups:
- Baseline [18F]MNI-1054: [18F]MNI-1054 up to 10 mCi, PET radiotracer injection, intravenously, prior to PET scan on Day -1 (Baseline scan).
- TAK-418 1.5 mg: TAK-418 1.5 mg, capsule, orally, once on Day 1 and up to 10 mCi of [18F]MNI-1054 PET radiotracer injection, intravenously, prior to each PET scans on Day 1, and either on Day 2 or 3 post-TAK-418 dose in the Treatment Period. All participants received [18F]MNI-1054 up to 10 mCi, injection, intravenously, prior to PET scan on Day -1 (Baseline scan).
- TAK-418 10 mg: TAK-418 10 mg, capsule, orally, once on Day 1 and up to 10 mCi of [18F]MNI-1054 PET radiotracer injection, intravenously, prior to each PET scans on Day 1, and either on Day 2 or 3 post-TAK-418 dose in the Treatment Period. All participants received [18F]MNI-1054 up to 10 mCi, injection, intravenously, prior to PET scan on Day -1 (Baseline scan).
- TAK-418 30 mg: TAK-418 30 mg, capsule, orally, once on Day 1 and up to 10 mCi of [18F]MNI-1054 PET radiotracer injection, intravenously, prior to each PET scans on Day 1, and either on Day 2 or 3 post-TAK-418 dose in the Treatment Period. All participants received [18F]MNI-1054 up to 10 mCi, injection, intravenously, prior to PET scan on Day -1 (Baseline scan).
Period: Baseline Scan (Day-1)
Arm/Group | Baseline [18F]MNI-1054 | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Started | 7 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Metabolites of [18F]MNI-1054 could not be analyzed | 1 | 0 | 0 | 0
Period: Treatment Period (Day 1 Through Day 2-3)
Arm/Group | Baseline [18F]MNI-1054 | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Started | 0 | 2 (Eligible participants from Baseline Period who received 10 mCi of [18F]MNI-1054 on Day -1.) | 2 (Eligible participants from Baseline Period who received 10 mCi of [18F]MNI-1054 on Day -1.) | 2 (Eligible participants from Baseline Period who received 10 mCi of [18F]MNI-1054 on Day -1.)
Completed | 0 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all enrolled participants who received at least 1 dose of [18F]MNI-1054 or TAK-418.
Arm/Group | Baseline [18F]MNI-1054
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 3
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.81 (2.594)

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Estimates of Binding of [18F]MNI-1054 Based on PET Radiotracer Kinetic Models At Baseline Scan on Day -1
Description: Enzyme binding parameter [Ki] was obtained from irreversible 2-tissue compartment model (mL/cm^3/min). Data is reported for the following brain regions: cerebellum, frontal lobe, hippocampus, occipital Lobe, pons, and striatum. Here, mL/cm^3/min signifies 'milliliter per cubic centimeter per minute'.
Time Frame: Day -1
Population: The pharmacodynamics (PD) set included all participants who received TAK-418 and have at least 1 analyzable PET Scan following TAK-418.
Measure: Mean (Standard Deviation); unit: mL/cm^3/min
Arm/Group | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Number analyzed (Participants) | 2 | 2 | 2
mL/cm^3/min
  Cerebellum | 0.03405 (0.002192) | 0.03515 (0.005869) | 0.03560 (0.003394)
  Frontal Lobe | 0.01930 (0.004525) | 0.02070 (0.004384) | 0.02140 (0.002263)
  Hippocampus | 0.01900 (0.000141) | 0.01935 (0.005303) | 0.01960 (0.001414)
  Occipital Lobe | 0.02140 (0.002404) | 0.02225 (0.003606) | 0.02365 (0.002616)
  Pons | 0.01685 (0.000071) | 0.01855 (0.004313) | 0.01870 (0.004667)
  Striatum | 0.01575 (0.004031) | 0.01930 (0.004950) | 0.01995 (0.003323)

2. Primary Outcome: Quantitative Estimates of Binding of [18F]MNI-1054 Based on PET Radiotracer Kinetic Models on Day 1
Description: as for outcome 1
Time Frame: Day 1
Population: The PD set included all participants who received TAK-418 and have at least 1 analyzable PET Scan following TAK-418.
Measure: Mean (Standard Deviation); unit: mL/cm^3/min
Arm/Group | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Number analyzed (Participants) | 2 | 2 | 2
mL/cm^3/min
  Cerebellum | 0.01020 (0.003536) | 0.00405 (0.000495) | 0.00760 (0.000849)
  Frontal Lobe | 0.01295 (0.001768) | 0.00980 (0.001697) | 0.01435 (0.002333)
  Hippocampus | 0.01260 (0.000990) | 0.00635 (0.004031) | 0.01240 (0.000000)
  Occipital Lobe | 0.01245 (0.002758) | 0.00910 (0.000990) | 0.01430 (0.001556)
  Pons | 0.01265 (0.006718) | 0.00970 (0.000707) | 0.01515 (0.000212)
  Striatum | 0.01185 (0.002192) | 0.00785 (0.000495) | 0.01365 (0.000071)

3. Primary Outcome: Quantitative Estimates of Binding of [18F]MNI-1054 Based on PET Radiotracer Kinetic Models on Day 2
Description: as for outcome 1
Time Frame: Day 2
Population: The PD set included all participants who received TAK-418 and have at least 1 analyzable PET Scan following TAK-418.
Measure: Mean (Standard Deviation); unit: mL/cm^3/min
Arm/Group | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Number analyzed (Participants) | 2 | 2 | 2
mL/cm^3/min
  Cerebellum | 0.01865 (0.004455) | 0.00875 (0.001485) | 0.00690 (0.000566)
  Frontal Lobe | 0.01610 (0.003111) | 0.01020 (0.001838) | 0.01130 (0.002404)
  Hippocampus | 0.01650 (0.003960) | 0.00865 (0.001061) | 0.01015 (0.000919)
  Occipital Lobe | 0.01665 (0.003889) | 0.01045 (0.002192) | 0.01180 (0.001980)
  Pons | 0.01265 (0.004738) | 0.01045 (0.002475) | 0.00985 (0.000636)
  Striatum | 0.01410 (0.004667) | 0.00915 (0.003182) | 0.00965 (0.001344)

4. Primary Outcome: Percent Enzyme Occupancy Based on Quantitative Estimates of Binding for TAK-418 on Day 1
Description: Lysine-Specific Demethylase 1A (LSD1) enzyme occupancy (%) in region of interest (ROI) after a single dose of TAK-418 was obtained from the baseline and postdose Ki values as follows: occupancy (1st postdose) = 100*(Ki [baseline] - Ki [1st postdose]) / Ki (baseline). Data is reported for following brain regions: cerebellum, frontal lobe, hippocampus, occipital Lobe, pons, and striatum.
Time Frame: Day 1
Population: The PD set included all participants who received TAK-418 and have at least 1 analyzable PET Scan following TAK-418.
Measure: Mean (Standard Deviation); unit: percentage of occupancy
Arm/Group | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Number analyzed (Participants) | 2 | 2 | 2
percentage of occupancy
  Cerebellum | 68.5 (10.61) | 87.0 (1.41) | 79.5 (2.12)
  Frontal Lobe | 19.5 (10.61) | 44.0 (9.90) | 38.0 (9.90)
  Hippocampus | 33.0 (5.66) | 59.5 (26.16) | 40.0 (0.00)
  Occipital Lobe | 37.0 (14.14) | 54.5 (4.95) | 43.5 (6.36)
  Pons | 25.0 (39.60) | 37.5 (4.95) | 31.0 (1.41)
  Striatum | 8.0 (16.97) | 50.5 (3.54) | 39.0 (0.00)

5. Primary Outcome: Percent Enzyme Occupancy Based on Quantitative Estimates of Binding for TAK-418 on Day 2
Description: LSD1 enzyme occupancy (%) in ROI after a single dose of TAK-418 was obtained from the baseline and postdose Ki values as follows: occupancy (2nd postdose) = 100*(Ki [baseline] - Ki [2nd postdose]) / Ki (baseline). Data is reported for following brain regions: cerebellum, frontal lobe, hippocampus, occipital Lobe, pons, and striatum.
Time Frame: Day 2
Population: The PD set included all participants who received TAK-418 and have at least 1 analyzable PET Scan following TAK-418.
Measure: Mean (Standard Deviation); unit: percentage of occupancy
Arm/Group | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Number analyzed (Participants) | 2 | 2 | 2
percentage of occupancy
  Cerebellum | 42.5 (13.44) | 71.5 (4.95) | 82.0 (1.41)
  Frontal Lobe | 0.5 (19.09) | 42.0 (9.90) | 51.0 (9.90)
  Hippocampus | 13.0 (21.21) | 44.5 (6.36) | 50.5 (4.95)
  Occipital Lobe | 16.0 (19.80) | 47.0 (11.31) | 53.5 (7.78)
  Pons | 25.0 (28.28) | 32.5 (16.26) | 55.0 (2.83)
  Striatum | -9.0 (35.36) | 42.0 (19.80) | 56.5 (6.36)

6. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-418
Time Frame: Day 1: pre-dose and at multiple time points (up to 3 hours) post-dose, immediately before and after the Day 1 PET scan, and within 30 minutes before and 30 minutes after Day 2 or 3 PET scan
Population: The pharmacokinetic (PK) set included all participants from the safety set who received TAK-418 and had at least 1 measurable plasma concentration for TAK-418.
Measure: Median (Full Range); unit: nanogram per milliliter (ng/mL)
Arm/Group | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Number analyzed (Participants) | 2 | 2 | 2
nanogram per milliliter (ng/mL) | 4.420 [4.23 to 4.61] | 43.80 [36.7 to 50.9] | 130.5 [127 to 134]

7. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve (AUC) From Time 0 to Time of the Last Quantifiable Concentration for TAK-418
Time Frame: as for outcome 6
Population: The PK set included all participants from the safety set who received TAK-418 and had at least 1 measurable plasma concentration for TAK-418.
Measure: Median (Full Range); unit: hour*nanogram per milliliter(h*ng/mL)
Arm/Group | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Number analyzed (Participants) | 2 | 2 | 2
hour*nanogram per milliliter(h*ng/mL) | 22.40 [20.8 to 24.0] | 227.5 [223 to 232] | 812.0 [718 to 906]

8. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-418
Time Frame: as for outcome 6
Population: The PK set included all participants from the safety set who received TAK-418 and had at least 1 measurable plasma concentration for TAK-418. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Number analyzed (Participants) | 1 | 2 | 2
h*ng/mL | 25.60 [25.6 to 25.6] | 230.0 [225 to 235] | 817.0 [721 to 913]

9. Secondary Outcome: ED50 PET Enzyme Occupancy
Description: The relationship between PET enzyme occupancy and TAK-418 dose level was investigated using an Emax model containing the regression parameters maximal target occupancy (Emax) and dose that gives 50 percent (%) of Emax (ED50). ED50 values are reported for following brain regions: cerebellum, frontal lobe, hippocampus, occipital Lobe, pons, and striatum. The data tabulated are the estimated value and confidence intervals of the ED50 value derived from an Emax model fit across all data points from all arms. ED50 is the dose at which 50% enzyme occupancy is expected.
Time Frame: Days 1 to 2
Population: The PD set included all participants who received TAK-418 and have at least 1 analyzable PET Scan following TAK-418
Measure: Mean (95% Confidence Interval); unit: milligram (mg)
Groups:
- TAK-418: TAK-418 1.5 mg, 10 mg, or 30 mg capsules, orally, once on Day 1 and up to 10 mCi of [18F]MNI-1054 PET radiotracer injection, intravenously, prior to each PET scans on Day 1, and either on Day 2 or 3 post-TAK-418 dose. All participants received [18F]MNI-1054 up to 10 mCi, injection, intravenously, prior to PET scan on Day -1 (Baseline scan).
Arm/Group | TAK-418
Number analyzed (Participants) | 6
milligram (mg)
  Cerebellum | 0.756 [0.288 to 1.224]
  Frontal Lobe | 4.328 [0.129 to 8.527]
  Hippocampus | 1.639 [-0.098 to 3.377]
  Occipital Lobe | 1.416 [0.141 to 2.690]
  Pons | 1.112 [-0.976 to 3.200]
  Striatum | 7.496 [-2.050 to 17.04]

10. Secondary Outcome: Number of Participants Reporting One or More Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose of [18F]MNI-1054 radiotracer injection up to Day 14
Population: The safety set included all enrolled participants who received at least 1 dose of [18F]MNI-1054 or TAK-418
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline [18F]MNI-1054 | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Number analyzed (Participants) | 7 | 2 | 2 | 2
Participants
  AEs | 1 | 0 | 1 | 2
  SAEs | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Values
Time Frame: From first dose of [18F]MNI-1054 radiotracer injection up to Day 14
Population: The safety set included all enrolled participants who received at least 1 dose of [18F]MNI-1054 or TAK-418
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline [18F]MNI-1054 | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Number analyzed (Participants) | 7 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Vital Signs
Time Frame: From first dose of [18F]MNI-1054 radiotracer injection up to Day 14
Population: The safety set included all enrolled participants who received at least 1 dose of [18F]MNI-1054 or TAK-418.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline [18F]MNI-1054 | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
Number analyzed (Participants) | 7 | 2 | 2 | 2
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first administration of [18F]MNI-1054 radiotracer injection until the Day 14
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Baseline [18F]MNI-1054 | TAK-418 1.5 mg | TAK-418 10 mg | TAK-418 30 mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/7 | 0/2 | 1/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baseline [18F]MNI-1054 (N=7) | TAK-418 1.5 mg (N=2) | TAK-418 10 mg (N=2) | TAK-418 30 mg (N=2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT04202497/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT04202497/SAP_001.pdf